CLINICAL TRIAL: NCT05985759
Title: Comparative Evaluation of the Effect of 970 nm Diode Laser With or Without N Acetyl Cysteine on Post Operative Pain After Endodontic Treatment in Teeth With Symptomatic Apical Periodontitis: a Randomized Clinical Trial
Brief Title: Comparative Evaluation of the Effect of 970 nm Diode Laser With or Without N Acetyl Cysteine on Post Operative Pain After Endodontic Treatment in Teeth With Symptomatic Apical Periodontiti
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bapuji Dental College & Hospital Davengere Karnataka (Other)
Responsible Party: Principal Investigator, JOE PAUL UMBAVU, post graduate student, Bapuji Dental College & Hospital Davengere Karnataka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECR1652InstKA2022/230506010
Record Dates: First submitted 2023-07-21; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Evaluation of Post Endodontic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 970nm diode laser (No Intervention)
- N acetyle cystiene (Experimental)
  Interventions: Drug: N acetyle cystiene
- calcium hydroxide (No Intervention)

INTERVENTIONS:
Drug: N acetyle cystiene — N acetyle cystien is administerd due to its antibacterial action and anti inflamatory action
  Arms: N acetyle cystiene

SUMMARY:
One of the most important aspect of endodontic treatment is management of postoperative pain management . Post operative pain after endodontic treatment is a frequent complication. frequency of post operative pain is between 3% to 58% .

Post operative pain could also occur as a result of inadequate instrumentation, extrusion of irrigation solutions, extrusion of intra-canal dressing, traumatic occlusion, missed canals, preoperative pain, periapical pathosis and extrusion of apical debris. Furthermore, instrument choice might also play an important role. The apical extrusion of infected debris during chemo-mechanical instrumentation of root canals might exacerbate the inflammatory response and cause peri-radicular inflammation.

The use of diode lasers, in addition to conventional endodontic therapy, has recently been proposed in RCT Various researchers have observed effective disinfection of the root canal by diode laser irradiation Due to the large water transmission capacities of diode lasers (810, 940 and 980-nm wavelengths), they can reach bacteria in deeper layers of dentinal tubules(3) Schoop et al. reported that using a 980-nm diode laser resulted in changes in dentinal surfaces and an increased bactericidal effect.

Other studies noted that laser irradiation decreases PP after RCT Over the years, studies have focused on identifying molecular mediators of inflammation induction, such as cytokines and chemokines in apical periodontitis. It was widely accepted that the loss of pro-inflammatory mediators was the 'turn off' signal of inflammation, ending subsequent responses passively.

Karapinar et al N-acetylcysteine (NAC) has been proposed as a potential alternative therapeutic agent in root canal treatment. NAC is an antioxidant mucolytic agent derivative of the amino acid L cysteine. As the precursor of glutathione, NAC can incorporate into cells and neutralize oxygen-derived free radicals (ROS), diminishing the cumulative effects of oxidative stress Previous studies have demonstrated the antimicrobial properties of NAC against several biofilm phenotypes, including oral pathogens such as Enterococcus faecalis, which is often found in endodontic infections. Moreover, NAC has been reported to exert anti-inflammatory activity by inhibiting the expression of lipopolysaccharide-induced inflammatory mediators.

Another study showed that the antibacterial effect of NAC is higher than that of NaOCl and CHX. More specifically, 200 mg/ ml solution of NAC was found to be more efficient than 5.25% NaOCl and 2% CHX in killing E. faecalis and S. mutant bacteria.(5) NAC exerts anti-inflammatory activity through its ability to inhibit the expression and release of a variety of proinflammatory cytokines. NAC can be a substitute for ibuprofen for post-endodontic pain. All these findings provide support for a superior potential for NAC in endodontic treatment.(6) Due to the scarcity of information on the effect of NAC as an intracanal medication, and the lack of systematic review on the same, this study aimed to compare and evaluate the post-operative pain when 970nm diode laser used with or without N acetyl cysteine as intracanal medicament

RESEARCH QUESTION : Will there be a difference in the postoperative pain after Endodontic treatment of mandibular molars with symptomatic apical periodontitis using 970nm diode laser with or without N acetyl cysteine ?

RESEARCH HYPOTHESIS (H1): There will be a difference in the postoperative pain after Endodontic treatment of mandibular molars with symptomatic apical periodontitis using 970nm diode laser with or without N acetyl cysteine

NULL HYPOTHESIS (H0): There will be no difference in the postoperative pain after Endodontic treatment of mandibular molars with symptomatic apical periodontitis using 970nm diode laser with or without N acetyl cysteine

DETAILED DESCRIPTION:
1. To assess the postoperative pain after Endodontic treatment of mandibular molars with symptomatic apical periodontitis using N acetyl cysteine as intracanal medicament
2. To assess the postoperative pain after Endodontic treatment of mandibular molars with symptomatic apical periodontitis using 970nm diode laser .
3. To assess the postoperative pain after Endodontic treatment of mandibular molars with symptomatic apical periodontitis using 970nm diode laser with N acetyl cysteine .
4. To compare the incidence of postoperative pain after endodontic treatment of mandibular molar with symptomatic apical periodontitis using N acetyl cysteine , 970nm diode laser , 970nm diode laser and N acetyl cysteine as intracanal medicament

7. MATERIALS AND METHODS: 7.1 TYPE OF STUDY: An in vivo study 7.2 SOURCE: The study will be performed on mandibular molar. Study is to be conducted in Dept. of Conservative Dentistry and Endodontics, BDCH, Davangere

7.3 Materials and Equipment

* 4 round bur ( Mani ,Japan ) Endo Z bur (Dentsply Sirona , India)
* 10, #15 K files of 21mm length (MANI) Protaper gold (DENTSPLY SIRONA) of 21mm length Disposable syringes (BD Glide) Side vented needle (neoendo) Beakers 0.9% Normal saline (INFUTEC NS) Airotor handpiece (Rotomax) Canalpro cl2i endomotor (Coltene ,India) Apex locater (j morita root zx) 17% EDTA solution (DENTAL AVENUE) 2.5% NaOCl solution (SDFCL) N acetyl cysteine (Sigma Aldrich , Merck KGaA, Darmstadt, Germany) Sirolaser blue (Sirolaser blue , Dentsply Maillefer, Ballaigues, Switzerland) Cavit (Cavit-G; 3 M ESPE, St Paul, MN) EQUIPMENT

  * X ray PSP scanner (PSP -SOREDEX DIGORA Optime) 7.2 Method of collection of data (including sampling procedure, if any): Simple random

METHODOLOGY Mandibular block anesthesia performed using local anesthetics solution 1.8ml 2% lidocaine with 1:80000 epinephrine. The procedure started after lip numbness was achieved. Occlusal reduction will be done followed by straight-line access cavity and the procedure was completed under rubber dam isolation. The working length was determined using an electronic apex locator (J morita), and Endomotor (Canalpro cl2i ,Coltene ,India) , Protaper gold (Dentsply Maillefer, Ballaigues, Switzerland) was used according to the manufacturer's instructions for cleaning and shaping .

A size 10 K-file was used to maintain apical patency, 2 mL 2.5% sodium hypochlorite was used between in-and-out pecking motions, and After instrumentation, The needle was advanced to a depth of 2-3 mm short of WL and the canal will be irrigated with 3 mL of 2.5% NaOCl. Final irrigation will be done with 5 mL of 17% EDTA for 1 min followed by a final rinse with 5ml of saline.

Randomization After that, patients were randomly assigned to one of the three groups based on the post operative therapy

ROOT CANAL INSTRUMENTATION

The patients will be randomly divided into 3 groups containing teeth in each group namely:

GROUP I(n=20): N acetyl cysteine GROUP II(n=20) : 970 nm diode laser Group II(n=20): 970 nm diode laser + N acetyl cysteine

Group I :

After the canals are dried with paper point N acetyl cysteine paste was applied as intra-canal medicament , and the access cavity was sealed using a temporary restorative material

GROUP II:

The final irrigation was performed , after the canals were dried with paper-points. During the laser treatment, both the operator and patient wore protective eyewear. Laser irradiation was applied using a 970-nm diode laser (Sirolaser blue , Dentsply Maillefer, Ballaigues, Switzerland) coupled with a 200-μm optical fibre. The settings were as follows: output power of 1.5 W in the pulsed mode irradiation for 10 s, followed by a 10-s pause, which comprised one cycle. This cycle was applied four times to each root canal. The power used was 1.5 W with a low frequency of 15 Hz. The optical fibre tip (length of 25 mm) was inserted at the working length. The root canals were then slowly (at a speed of 2 mm/s) irradiated from the apical to coronal using a continuous circling movement touching the dentinal walls in one cycle for each power. and the access cavity was sealed using a temporary restorative material.

GROUP III:

The final irrigation was performed as in the control group, and the canals were dried with paper points. During the laser treatment, both the operator and patient wore protective eyewear. Laser irradiation was applied using a 970-nm diode laser (sirolaser blue Dentsply Maillefer, Ballaigues, Switzerland ) coupled with a 200-μm optical fibre .The settings were as follows: power of 1.5 W and in the pulsed mode , irradiation for 10 s, followed by a 10-s pause, which comprised one cycle. This cycle was applied four times to each root canal. The power used was 1.5 W with a low frequency of 15 Hz. The optical fibre tip (length of 25 mm) was inserted at the working length. The root canals were then slowly (at a speed of 2 mm/s) irradiated from the apical to coronal using a continuous circling movement touching the dentinal walls in one cycle for each power.

Following the irradiation procedure, N acetyl cysteine paste was applied as intra-canal medicament , and the access cavity was sealed using a temporary restorative material, as in the control group

Subsequently, a temporary restorative material (Cavit-G; 3 M ESPE, St Paul, MN) was used to seal the access cavity.

At the time of the first visit, all the patients were given a VAS to rate their PP. A second appointment was scheduled for 7 d later. All patients who met the final inclusion criteria were given a pain chart to be completed to record the incidence of pain (yes/no), level of posttreatment pain and duration of pain (days).

The following variables were recorded:

1. Age
2. Sex
3. Tooth number
4. Number of canals

6. Preoperative pain on the VAS 7. Preoperative and postoperative percussion pain levels (on the 7th day) on the VAS 8. Pain level on the 8 hr ,24 hr, 48hr , 72hr & 7 day 11. Analgesic intake after the procedure

At the second appointment, the ICM was removed from the root canals with final irrigation and using an F3/F2 file. The root canals were then obturated using the cold lateral condensation method with gutta-percha cones and AH Plus sealer (Dentsply Maillefer, Ballaigues, Switzerland). The coronal restoration was finished using a resin composite (Filtek Z250, 3 M ESPE, St. Paul, MN).

ELIGIBILITY:
Inclusion Criteria:• Patients with mandibular molar with symptomatic apical periodontitis

* Periapical index up to 3 or 4.(8)
* Patient older than 18 to 60 years
* Spontaneous pain <3mm
* Percussion pain <3mm
* healthy induvidual

Exclusion Criteria:

* • Periodontal probing greater than 3mm

  * Previous root canal treatment
  * Swelling / sinus tract
  * Sever periodontal disease
  * Antibiotic use within last 5 days
  * Systemic disorders
  * Pregnancy and lactation
  * Traumatic occlusion
  * Severe crown destruction preventing rubber dam isolation
  * Presence of other teeth requiring RCT

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
modified visual analog scale | 7 days
  evaluation of post endodontic pain

CONTACTS AND LOCATIONS:
Locations (1):
- Bapuji Dental College and Hospital , Davangere, Davangere, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided